CLINICAL TRIAL: NCT04658797
Title: Clinical Evaluation on Using Personal Face Masks With Spectacles Versus Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C20-688 (EX-MKTG-120)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Single Vision Spectacle for Vision correction (Active Comparator): Single Vision Spectacle
  Interventions: Device: Single Vision Spectacle for Vision Correction; Other: Personal Facemask
- somofilcon A Daily disposable contact lenses (Experimental): Daily disposable contact lenses
  Interventions: Device: somofilcon A Daily Disposable Contact Lens; Other: Personal Facemask

INTERVENTIONS:
Device: somofilcon A Daily Disposable Contact Lens — Daily Disposable Contact Lens
  Arms: somofilcon A Daily disposable contact lenses
Device: Single Vision Spectacle for Vision Correction — Single Vision Spectacle
  Arms: Single Vision Spectacle for Vision correction
Other: Personal Facemask — Personal Facemask

SUMMARY:
The aim of this study was to explore satisfaction with vision correction and ease of use of PFM (Personal Face Masks) in a group of spectacle wearers who were randomised to continue wearing spectacles or be fitted with daily disposable contact lenses.

DETAILED DESCRIPTION:
This was a two arm parallel-group, randomised study. Subjects wearing single vision spectacles were recruited to participate in the study. Subjects were randomised to either continue to use their spectacles or to be fitted with the study daily disposable (DD) contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. They are aged between 18 and 40 years.
2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They are a 'neophyte' (i.e. someone who has not worn contact lenses previously, with the exception for the purposes of a trial fitting).
5. They have a contact lens spherical prescription between +8.00D and -10.00D (inclusive) based on the ocular refraction.
6. They have a cylindrical correction of -0.75DC or less in each eye based on the ocular refraction.
7. They own and habitually wear single vision spectacles.
8. They are willing to be fitted with contact lenses and understand they may be randomised to either group.
9. They are willing to wear the contact lenses (if relevant) or spectacles for at least 8 hours per day, 5 days per week.
10. They are able to wear the supplied surgical masks for the majority of time that they need to wear PFM and will wear the PFM for at least one hour a day for at least four days per week.
11. They can attain at least 0.20 logMAR distance high contrast visual acuity in each eye with the study lenses (if relevant) or spectacles.
12. They agree to not participate in other clinical research while enrolled on this study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens
2. wear.
3. They have a systemic disorder which would normally contra-indicate contact lens wear.
4. They are using any topical medication such as eye drops or ointment.
5. They have had cataract surgery.
6. They have had corneal refractive surgery.
7. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
8. They are pregnant or breastfeeding.
9. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
10. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
11. They require significant ocular/face personal protective equipment beyond a personal face mask.
12. They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.
13. They have spectacles which are not within ±0.50D of their refractive error.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codina, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Vision Spectacle for Vision Correction: Subjects were randomized to wear Single Vision Spectacle for Vision Correction: Single Vision Spectacle along with personal Facemask.
- Somofilcon A Daily Disposable Contact Lenses: Subjects were randomized to wear somofilcon A Daily Disposable Contact Lens along with personal Facemask.
Period: Overall Study
Arm/Group | Single Vision Spectacle for Vision Correction | Somofilcon A Daily Disposable Contact Lenses
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Vision Spectacle for Vision Correction | Somofilcon A Daily Disposable Contact Lenses | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (5.3) | 27.4 (5.8) | 26.5 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - High Contrast
Description: Visual Acuity under high contrast was measured using logMAR Visual Acuity Chart
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
logMAR | -0.06 (0.07) | -0.07 (0.05)

2. Primary Outcome: Visual Acuity - Low Contrast
Description: Visual Acuity under low contrast was measured using logMAR Visual Acuity Chart
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
logMAR | 0.20 (0.10) | 0.21 (0.07)

3. Primary Outcome: Visual Acuity - High Contrast
Description: Visual Acuity under high contrast was measured using logMAR Visual Acuity Chart
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
logMAR | -0.08 (0.08) | -0.08 (0.05)

4. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Breathability
Description: Subjective response on facemask usability questionnaire - Breathability assessed on a 5 point scale (1- very unsatisfactory, 2- Unsatisfactory, 3- Average, 4- Satisfactory, 5- Very Satisfactory)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very Satisfactory | 1 | 2
  Satisfactory | 4 | 5
  Average | 5 | 6
  Unsatisfactory | 4 | 2
  very unsatisfactory | 1 | 0

5. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Breathability
Description: as for outcome 4
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very Satisfactory | 5 | 1
  Satisfactory | 5 | 5
  Average | 5 | 6
  Unsatisfactory | 0 | 2
  very unsatisfactory | 0 | 1

6. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Heat
Description: Subjective response on facemask usability questionnaire - Heat assessed on a 5 point scale (1- very unsatisfactory, 2- Unsatisfactory, 3- Average, 4- Satisfactory, 5- Very Satisfactory)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very Satisfactory | 1 | 0
  Satisfactory | 2 | 6
  Average | 3 | 4
  Unsatisfactory | 8 | 4
  very unsatisfactory | 1 | 1

7. Primary Outcome: Subjective Response on Facemask Usability Questionnaire -Heat
Description: as for outcome 6
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very Satisfactory | 3 | 1
  Satisfactory | 6 | 2
  Average | 4 | 4
  Unsatisfactory | 2 | 7
  very unsatisfactory | 0 | 1

8. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Tightness
Description: Subjective response on facemask usability questionnaire - Tightness assessed on a 5 point scale (1- very unsatisfactory, 2- Unsatisfactory, 3- Average, 4- Satisfactory, 5- Very Satisfactory)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 2 | 2
  Satisfactory | 7 | 7
  Average | 4 | 5
  Unsatisfactory | 2 | 1
  Very unsatisfactory | 0 | 0

9. Primary Outcome: Subjective Response on Facemask Usability Questionnaire -Tightness
Description: as for outcome 8
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 4 | 0
  Satisfactory | 7 | 10
  Average | 3 | 5
  Unsatisfactory | 1 | 0
  Very unsatisfactory | 0 | 0

10. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Ease in Talking
Description: Subjective response on facemask usability questionnaire - Ease in Talking assessed on a 5 point scale (1- very unsatisfactory, 2- Unsatisfactory, 3- Average, 4- Satisfactory, 5- Very Satisfactory)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 2 | 1
  Satisfactory | 3 | 6
  Average | 4 | 5
  Unsatisfactory | 5 | 3
  Very unsatisfactory | 1 | 0

11. Primary Outcome: Subjective Response on Facemask Usability Questionnaire -Ease in Talking
Description: as for outcome 10
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 3 | 1
  Satisfactory | 4 | 4
  Average | 4 | 6
  Unsatisfactory | 4 | 4
  Very unsatisfactory | 0 | 0

12. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Comfort on Ear Lobes
Description: Subjective response on facemask usability questionnaire - Comfort on ear lobes assessed on a 5 point scale (1- very unsatisfactory, 2- Unsatisfactory, 3- Average, 4- Satisfactory, 5- Very Satisfactory)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 8 | 3
  Satisfactory | 2 | 7
  Average | 1 | 2
  Unsatisfactory | 3 | 3
  Very unsatisfactory | 1 | 0

13. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Comfort on Ear Lobes
Description: as for outcome 12
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 6 | 4
  Satisfactory | 5 | 6
  Average | 3 | 2
  Unsatisfactory | 1 | 3
  Very unsatisfactory | 0 | 0

14. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Overall Comfort
Description: Subjective response on facemask usability questionnaire - Overall Comfort assessed on a 5 point scale (1- very unsatisfactory, 2- Unsatisfactory, 3- Average, 4- Satisfactory, 5- Very Satisfactory)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 0 | 0
  Satisfactory | 2 | 5
  Average | 8 | 10
  Unsatisfactory | 4 | 0
  Very unsatisfactory | 1 | 0

15. Primary Outcome: Subjective Response on Facemask Usability Questionnaire - Overall Comfort
Description: as for outcome 14
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very satisfactory | 3 | 0
  Satisfactory | 6 | 4
  Average | 5 | 7
  Unsatisfactory | 1 | 2
  Very unsatisfactory | 0 | 2

16. Primary Outcome: Difficulty in Walking When Using Wearing Vision Correction and Facemask
Description: Difficulty in walking when using wearing vision correction and facemask assessed on a scale of 1-5 (1- very difficult, 2- difficult, 3- Neutral, 4, Easy, 5- Very Easy).
Time Frame: Baseline
Population: One subject from somofilcon A Daily disposable contact lenses didn't answer questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 14 | 15
Participants
  Very easy | 1 | 3
  Easy | 3 | 1
  Neutral | 2 | 4
  Difficult | 4 | 6
  Very difficult | 4 | 1

17. Primary Outcome: Difficulty in Walking When Using Wearing Vision Correction and Facemask
Description: as for outcome 16
Time Frame: 2 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very easy | 11 | 3
  Easy | 4 | 3
  Neutral | 0 | 3
  Difficult | 0 | 5
  Very difficult | 0 | 1

18. Primary Outcome: Difficulty in Driving When Using Wearing Vision Correction and Facemask
Description: Difficulty in driving when using wearing vision correction and facemask assessed on a scale of 1-5 (1- very difficult, 2- difficult, 3- Neutral, 4, Easy, 5- Very Easy)
Time Frame: Baseline
Population: 10 subjects from somofilcon A Daily disposable contact lenses and 6 subjects from Single Vision Spectacle for Vision correction didn't drive with their face mask and didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 5 | 9
Participants
  Very easy | 0 | 0
  Easy | 0 | 1
  Neutral | 0 | 3
  Difficult | 2 | 2
  Very difficult | 3 | 3

19. Primary Outcome: Difficulty in Driving When Using Wearing Vision Correction and Facemask
Description: as for outcome 18
Time Frame: 2 weeks
Population: 11 subjects from somofilcon A Daily disposable contact lenses and 7 subjects from Single Vision Spectacle for Vision correction didn't drive with their face mask and didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 4 | 8
Participants
  Very Easy | 3 | 0
  Easy | 1 | 2
  Neutral | 0 | 2
  Difficult | 0 | 1
  Very Difficult | 0 | 3

20. Primary Outcome: Difficulty in Reading When Using Wearing Vision Correction and Facemask
Description: Difficulty in reading when using wearing vision correction and facemask assessed on a scale of 1-5 (1- very difficult, 2- difficult, 3- Neutral, 4, Easy, 5- Very Easy)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very easy | 1 | 2
  Easy | 1 | 2
  Neutral | 3 | 6
  Difficult | 7 | 4
  Very difficult | 3 | 1

21. Primary Outcome: Difficulty in Reading When Using Wearing Vision Correction and Facemask
Description: as for outcome 20
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very easy | 9 | 2
  Easy | 3 | 4
  Neutral | 3 | 3
  Difficult | 0 | 4
  Very difficult | 0 | 2

22. Primary Outcome: Difficulty in Working With a Computer When Using Wearing Vision Correction and Facemask
Description: Difficulty in working with a computer when using wearing vision correction and facemask assessed on a scale of 1-5 (1- very difficult, 2- difficult, 3- Neutral, 4, Easy, 5- Very Easy)
Time Frame: Baseline
Population: 3 subjects from somofilcon A Daily disposable contact lenses didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 12 | 15
Participants
  Very easy | 1 | 1
  Easy | 0 | 3
  Neutral | 1 | 4
  Difficult | 8 | 6
  Very difficult | 2 | 1

23. Primary Outcome: Difficulty in Working With a Computer When Using Wearing Vision Correction and Facemask
Description: as for outcome 22
Time Frame: 2 weeks
Population: 1 subject from somofilcon A Daily disposable contact lenses didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 14 | 15
Participants
  Very easy | 7 | 3
  Easy | 3 | 3
  Neutral | 3 | 3
  Difficult | 1 | 4
  Very difficult | 0 | 2

24. Primary Outcome: Difficulty in Exercising (Physical Activities) When Using Wearing Vision Correction and Facemask
Description: Difficulty in exercising (physical activities)when using wearing vision correction and facemask assessed on a scale of 1-5 (1- very difficult, 2- difficult, 3- Neutral, 4, Easy, 5- Very Easy)
Time Frame: Baseline
Population: 7 subjects from somofilcon A Daily disposable contact lenses and 4 subjects from Single Vision Spectacle for Vision correction didn't exercise with facemask and didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 8 | 11
Participants
  Very easy | 0 | 0
  Easy | 0 | 0
  Neutral | 0 | 0
  Difficult | 2 | 7
  Very difficult | 6 | 4

25. Primary Outcome: Difficulty in Exercising (Physical Activities) When Using Wearing Vision Correction and Facemask
Description: as for outcome 24
Time Frame: 2 weeks
Population: 2 subjects from somofilcon A Daily disposable contact lenses and 3 subjects from Single Vision Spectacle for Vision correction didn't exercise with facemask and didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 13 | 12
Participants
  Very Easy | 6 | 0
  Easy | 4 | 0
  Neutral | 3 | 0
  Difficult | 0 | 9
  Very Difficult | 0 | 3

26. Primary Outcome: Difficulty in Socializing When Using Wearing Vision Correction and Facemask
Description: Difficulty in socializing when using wearing vision correction and facemask assessed on a scale of 1-5 (1- very difficult, 2- difficult, 3- Neutral, 4, Easy, 5- Very Easy)
Time Frame: Baseline
Population: 1 subject from somofilcon A Daily disposable contact lenses didn't answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 14 | 15
Participants
  Very Easy | 0 | 2
  Easy | 2 | 2
  Difficult | 3 | 4
  Neutral | 4 | 5
  Very Difficult | 5 | 2

27. Primary Outcome: Difficulty in Socializing When Using Wearing Vision Correction and Facemask
Description: as for outcome 26
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Very easy | 6 | 2
  Easy | 5 | 2
  Difficult | 1 | 4
  Neutral | 3 | 5
  Very difficult | 0 | 2

28. Primary Outcome: Physical Safety Concerns When Wearing Your Vision Correction and Facemask
Description: Physical safety concerns when wearing your vision correction and facemask assessed on a scale of 1-5 (1- Extremely concerned, 2 - Moderately concerned, 3- Somewhat concerned, 4 -Slightly concerned, 5- Not at all concerned)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Not at all concerned | 6 | 9
  Slightly concerned | 1 | 3
  Somewhat concerned | 3 | 1
  Moderately concerned | 5 | 2
  Extremely concerned | 0 | 0

29. Primary Outcome: Physical Safety Concerns When Wearing Your Vision Correction and Facemask
Description: as for outcome 28
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Not at all concerned | 12 | 9
  Slightly concerned | 3 | 3
  Somewhat concerned | 0 | 1
  Moderately concerned | 0 | 1
  Extremely concerned | 0 | 1

30. Primary Outcome: Emotional Impact of Using the Facemask When Wearing Your Vision Correction
Description: Emotional impact of using the facemask when wearing your vision correction assessed on a scale of 1-5 (1- Severe, 2- Major, 3- Moderate, 4- Minor, 5- Insignificant)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Insignificant | 5 | 7
  Minor | 6 | 6
  Moderate | 3 | 2
  Major | 1 | 0
  Severe | 0 | 0

31. Primary Outcome: Emotional Impact of Using the Facemask When Wearing Your Vision Correction
Description: as for outcome 30
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Insignificant | 8 | 6
  Minor | 6 | 6
  Moderate | 1 | 3
  Major | 0 | 0
  Severe | 0 | 0

32. Primary Outcome: Impact of Using the Facemask on Your Personal Appearance When Wearing Your Vision Correction
Description: Impact of using the facemask on your personal appearance when wearing your vision correction assessed on a scale of 1-5 (1- Severe, 2- Major, 3- Moderate, 4- Minor, 5- Insignificant)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Insignificant | 5 | 2
  Minor | 3 | 6
  Moderate | 4 | 3
  Major | 3 | 3
  Severe | 0 | 1

33. Primary Outcome: Impact of Using the Facemask on Your Personal Appearance When Wearing Your Vision Correction
Description: as for outcome 32
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Somofilcon A Daily Disposable Contact Lenses | Single Vision Spectacle for Vision Correction
Number analyzed (Participants) | 15 | 15
Participants
  Insignificant | 7 | 3
  Minor | 6 | 8
  Moderate | 2 | 3
  Major | 0 | 0
  Severe | 0 | 1

ADVERSE EVENTS:
Time Frame: Subjects were randomized to wear single vision spectacle and somofilcon A daily disposable contact lenses along with personalized face masks - from dispense to 2 weeks visit - a total of two weeks.
Arm/Group | Single Vision Spectacle for Vision Correction | Somofilcon A Daily Disposable Contact Lenses
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT04658797/Prot_SAP_000.pdf